CLINICAL TRIAL: NCT01514578
Title: A Multi-Part, Randomized, Single-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous TRV130A in Healthy Adult Males
Brief Title: Single Ascending Dose Study of Intravenous TRV130A in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP130-1001
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: safety; tolerability; TRV130A
MeSH Terms: interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRV130A (Experimental)
  Interventions: Drug: TRV130A
- Dextrose in Water (Placebo Comparator)
  Interventions: Drug: Dextrose in Water

INTERVENTIONS:
Drug: TRV130A — Intravenous infusion of 1 hour duration
  Arms: TRV130A
Drug: Dextrose in Water — Intravenous infusion of 1 hour duration
  Arms: Dextrose in Water

SUMMARY:
This study will evaluate the safety, blood levels, and effects of TRV130A on pain perception and sedation in healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male 19 - 50 years of age
* Body weight >/= 50 kg
* Capable of giving written informed consent

Exclusion Criteria:

* Clinically significant disease or conditions that may place the subject at unacceptable risk as a participant in the study, or that may interfere with the safety, tolerability or pharmacodynamic evaluations in the study
* Laboratory tests positive for HIV, Hepatitis B virus surface antigen, or Hepatitis C virus antibody; elevations of aspartate aminotransferase or alanine aminotransferase; positive drug or alcohol test; positive urine test for cotinine
* Major surgery within 4 weeks of screening

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Baseline to 8 days after dose administration
Area under the plasma concentration versus time curve of TRV130A | Baseline to 24 hours after dose administration

SECONDARY OUTCOMES:
Effect of TRV130A on pain perception using cold pain test | Baseline to 3 hours after dose administration
Effect of TRV130A on pupil diameter | Baseline to 3 hours after dose administration
Effect of TRV130A on eye movements | Baseline to 3 hours after dose administration
  Using saccadic eye movement measurement
Effect of TRV130A on sedation | Baseline to 3 hours after dose administration
  Sedation evaluated by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David G. Soergel, MD, Study Director — Trevena Inc.; Alan S. Marion, MD, PhD, Principal Investigator — ICON Development Solutions
Locations (1):
- ICON Development Solutions, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Soergel DG, Subach RA, Sadler B, Connell J, Marion AS, Cowan CL, Violin JD, Lark MW. First clinical experience with TRV130: pharmacokinetics and pharmacodynamics in healthy volunteers. J Clin Pharmacol. 2014 Mar;54(3):351-7. doi: 10.1002/jcph.207. Epub 2014 Jan 28. PMID 24122908
- [Derived] Soergel DG, Subach RA, Cowan CL, Violin JD, Lark MW. First clinical experience with TRV027: pharmacokinetics and pharmacodynamics in healthy volunteers. J Clin Pharmacol. 2013 Sep;53(9):892-9. doi: 10.1002/jcph.111. Epub 2013 Jun 29. PMID 23813302